CLINICAL TRIAL: NCT01162343
Title: Delirium in the Emergency Department: Novel Screening
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Jin H. Han, MD, Vanderbilt University Medical Center
Other Study IDs: 081408
Record Dates: First submitted 2010-07-12; First posted 2010-07-14 (Estimated); Results first posted 2018-05-03 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Delirium
Keywords: Delirium, diagnosis, elderly, hospitalization
MeSH Terms: conditions — Delirium; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Older Emergency Department Patients: Patients who were 65 years or older from the emergency department were enrolled.

SUMMARY:
Delirium is an acute confusional state characterized by altered or fluctuating mental status, inattention, and either disorganized thinking or an altered level of consciousness. This form of organ dysfunction occurs in up to 10% of older emergency department (ED) patients and is associated with worsening mortality, prolonged hospital length of stay, higher health care costs, and accelerated functional and cognitive decline. Despite the negative consequences of delirium, the majority of cases are unrecognized by emergency physicians because it is not routinely screened for. In an effort to facilitate delirium screening, the investigators sought to validate three brief delirium assessments in the ED setting.

DETAILED DESCRIPTION:
Delirium is often missed because emergency physicians do not routinely screen for this diagnosis. Most delirium assessments can take up to 10 minutes to perform making them less likely to be incorporated into the routine physician assessment. Using brief (<2 minutes) and easy to use delirium assessments may ameliorate this quality of care issue. The Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) possesses these characteristics, but has only been validated in mechanically and non-mechanically ventilated intensive care unit patients. Recently, the investigators also developed the Brief Confusion Assessment Method (B-CAM) which is a modification of the CAM-ICU. The benefit is that it takes even less time than the CAM-ICU. The investigators also developed the Emergency Department Delirium Triage Screen (ED-DTS) designed to be highly sensitive and moderately specific delirium assessment for the nurse's triage assessment. It is hypothesized that a negative ED-DTS would rule out delirium, while a positive ED-DTS would require a more formal delirium assessment such as the CAM-ICU and B-CAM. These new delirium assessments require validation in older ED patients. As result, the investigators propose the following and the following specific aims:

Aim #1: To validate the B-CAM in older ED patients. The B-CAM will be performed by a clinical trials associate (CTA) and principal investigator in 200 ED patients that are > 65 years old. This instrument will be validated against a psychiatrist's Diagnostic and Statistical Manual of Mental Disorders, 4th. Edition Text Revision assessment as the reference standard.

Aim #2: To validate the CAM-ICU in older ED patients. The CAM-ICU will be performed by a clinical trials associate (CTA) and principal investigator in approximately 200 ED patients that are > 65 years old. This instrument will be validated against a psychiatrist's Diagnostic and Statistical Manual of Mental Disorders, 4th. Edition Text Revision assessment as the reference standard.

Aim #3: To validate the ED-DTS in older ED patients. The ED-DTS will be performed by a clinical trials associate (CTA) and principal investigator in 200 ED patients that are > 65 years old. This instrument will be validated against a psychiatrist's Diagnostic and Statistical Manual of Mental Disorders, 4th. Edition Text Revision assessment as the reference standard.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or greater
* In the Emergency Department for less than 12 hour at the time of enrollment

Exclusion Criteria:

* Severe mental retardation or dementia
* Baseline communication barriers such as aphasia, deafness, blindness, or who are unable to speak English
* Refusal of consent
* Previous enrollment
* Comatose
* Out of the hospital before the assessments are completed

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The participants will be those who are Vanderbilt University Emergency Department patients 65 years or older. There will be no selection bias in regards to race or gender. Only those who meet the inclusion/exclusion criteria will be considered for study inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 498 (Actual)
Dates: Start 2009-07; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jin H Han, MD, MSc, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: While 498 patients were enrolled, 92 were excluded from the final analysis because they did not receive a psychiatrist reference standard delirium assessment. As a result, 406 patients were included for the final analysis.
Period: Overall Study
Arm/Group | Older Emergency Department Patients
Started | 498
Completed | 406
Not Completed | 92
Not completed — Left ED prior to psychiatrist assessment | 80
Not completed — Refused psychiatrist assessment | 12

BASELINE CHARACTERISTICS:
Arm/Group | Older Emergency Department Patients
Number analyzed (Participants) | 406
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 73.5 [69 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 202
  Male | 204
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Non-white | 57
  Race: White | 349
Dementia documented in medical record [Count of Participants; unit: Participants] | 24
Charlson Comorbidity Index [Median (Inter-Quartile Range); unit: points on a scale] — Total range for the Charlson Comorbidity Index is 0 to 33. Higher values represent higher comorbidity burden.
  points on a scale | 2 [1 to 4]
Acute Physiology Score [Median (Inter-Quartile Range); unit: points on a scale] — Measured by APACHE II, a severity-of-disease classification system Higher values represent higher severity of illness (sicker). APACHE II score ranges from 0 to 71
  points on a scale | 2 [1 to 4]
Admitted to the hospital [Count of Participants; unit: Participants] | 294

OUTCOME MEASURES:

1. Primary Outcome: Delirium
Description: Delirium was diagnosed by a consultation-liaison psychiatrist assessment using Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria. The psychiatrists performed a battery of bedside cognitive tests, including (but not limited to) Clock Drawing Test, Luria hand sequencing task, and tests for verbal fluency. A focused neurological examination (i.e., screening for paraphasic errors, tremors, tone, asterixis, frontal release signs etc.,) and evaluation for affective lability, hallucinations, and level of alertness were also conducted routinely. Confrontational naming, proverb interpretation or similarities, and assessments for apraxias were performed at the discretion of the reference psychiatrists, especially if the diagnosis of delirium was inconclusive.
Time Frame: Within 3 hours of the study assessments.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Older Emergency Department Patients
Number analyzed (Participants) | 406
percent
  Research Assistant DTS Sensitivity | 98.0 [89.5 to 99.5]
  Research Assistant DTS Specificity | 56.2 [51.0 to 61.3]
  Physician DTS Sensitivity | 56.2 [51.0 to 61.3]
  Physician DTS Specificity | 54.8 [49.6 to 59.9]
  Research Assistant bCAM Sensitivity | 78.0 [64.8 to 87.2]
  Research Assistant bCAM Specificity | 96.9 [94.6 to 98.3]
  Physician bCAM Sensitivity | 84.0 [71.5 to 91.7]
  Physician bCAM Specificity | 95.8 [93.2 to 97.4]
  Research Assistant CAM-ICU Sensitivity | 68.0 [54.2 to 79.2]
  Research Assistant CAM-ICU Specificity | 98.6 [96.8 to 99.4]
  Physician CAM-ICU Sensitivity | 72.0 [58.3 to 82.5]
  Physician CAM-ICU Specificity | 98.6 [96.8 to 99.4]

ADVERSE EVENTS:
Arm/Group | Older Emergency Department Patients
All-Cause Mortality (participants affected / at risk) | 0/498
Serious Adverse Events (participants affected / at risk) | 0/498
Other Adverse Events (participants affected / at risk) | 0/498

LIMITATIONS AND CAVEATS:
This was a single center study and should be externally validated. Our findings cannot be generalized to those who are younger than 65 years old.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No